CLINICAL TRIAL: NCT05256706
Title: Evaluating the Impact of SomaSignal Tests on Medical Management and Change in Risk in Patients With Type 2 Diabetes at Higher Risk of Cardiovascular Disease
Brief Title: SomaSignal Tests on Medical Management and Change in Risk in Patients With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: SomaLogic, Inc. (Industry)
Responsible Party: Principal Investigator, Arshed A. Quyyumi, Professor of Medicine, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00003362
Record Dates: First submitted 2022-01-20; First posted 2022-02-25 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: cardiovascular risk
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- SomaSignal Informed Medical Management SSCVD (Experimental): Blood draw for SSCVD test at baseline and 6 months (±50 days). SomaSignal Cardiovascular Risk (SSCVD) results will be sent to the providers and participants approximately 2-4 weeks after testing.
  Interventions: Diagnostic Test: SomaSignal Informed Medical Management SSCVD
- Standard of Care (Uninformed Arm) (Active Comparator): Blood draw for SSCVD test at baseline and 6 months (±50 days). SomaSignal Cardiovascular Risk (SSCVD) results will not be provided to the provider or participant until the 6-month visit.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Diagnostic Test: SomaSignal Informed Medical Management SSCVD — For participants randomized to the Informed arm, the SSCVD test results will be provided to the participant's clinicians approximately 2-4 weeks after the baseline blood draw. Clinicians will discuss results with the participant and make adjustments to the care plan as needed based on the SSCVD test results within 50 days of receiving results. Clinicians may advise participants to (i) either change the doses of existing medications within existing guidelines, (ii) prescribe additional guideline-based medications, (iii) advise additional lifestyle interventions, or (iv) advise no change. This information will be documented in the case report forms. This test is neither intended to diagnose cardiovascular disease (CVD) nor replace the standard of care protocols for this disease. The physician should not rely solely on this information to make a decision on the best course of action for this patient.
  Other Names: SSCVD Informed
  Arms: SomaSignal Informed Medical Management SSCVD
Other: Standard of Care — Clinicians will provide the standard of care based on routine test results and without the SSCVD results. The SSCVD and SomaSignal Metabolic Factor Panel results from participants from both the baseline and 6-month period will be provided to the study team at the 6-month study visit. The SomaSignal Metabolic Factor tests include evaluation of Liver Fat, Glucose Tolerance, Kidney Function, Alcohol Impact, Cardiorespiratory Fitness/oxygen consumption (VO2) max, Resting Energy Rate, Body Fat Percentage, Visceral Fat, and Lean Body Mass. Any recommendations made to the participant by the physicians, based on obtaining the aforementioned test results will be collected.
  Other Names: Uninformed Arm
  Arms: Standard of Care (Uninformed Arm)

SUMMARY:
Despite the development of novel treatments, cardiovascular disease (CVD) remains the leading cause of death and disability. It has been observed in clinical practice, that the use of novel glycemia-lowering therapies with cardioprotective features remains profoundly low despite proven efficacy. It has been proposed that such low uptake is more related to insurance type and coverage than to risk assessment. While it can be easy to blame prescribing deficiencies on complacent physicians and/or over-frugal payors, SomaLogic believes there is more likely to be a fundamental problem with the cost and risk-effective allocation of such therapies, which are neither low in cost nor free of adverse events. As current clinical trials and guidelines tend to "bundle" participants together, there is an absence of individualized assessment of residual cardiovascular risk. This leads to physicians, participants, and payors being relatively uninformed as to the need for and/or likely benefits of such therapies in an individual. Simply giving every eligible participant a drug regardless of residual risk would be unaffordable and would create adverse effects and costs for people at low residual risk who might not actually benefit from the drugs.

To resolve this lack of precision in risk assessment, SomaLogic has performed the largest ever proteomic program to date with over 36,000 samples from 26,000 participants in eleven clinical studies, for a total of over 180,000,000 protein measurements, to develop and validate a surrogate proteomic endpoint for cardiovascular outcomes. The SomaSignal Cardiovascular Risk (SSCVR) test, a 27-protein model encompassing ten biological systems.

DETAILED DESCRIPTION:
This study is being done to evaluate the use of a new test for the management and treatment of patients who are at high risk of heart disease. The test, called a "SomaSignal Test", makes use of personalized proteomics. "Proteomes" refer to a set of proteins produced in the body. Proteins can affect the function of our bodies and can regulate disease, behavior, and drug treatments. The research team's hypothesis is that the SomaSignal Test can study these proteins and provide results that can help in the management of heart disease.

Potential benefits include increased participant engagement and satisfaction from increased personalized medical knowledge and improved participant outcomes through personalized risk stratification, more precise clinical care, and improvements in the triage of medical interventions and education. There may be improved health outcomes in the subset of participants who have a residual risk based on the SomaSignal Test test that they were previously unaware of, and who may receive treatment with a drug or additional lifestyle intervention they were previously eligible for but were not undertaking at the start of the study.

All participating providers will be provided education and training on SomaSignal testing including how to interpret and educate participants on the results. There will be two study visits. Participants will be randomized into one of 2 arms. Blood samples and information collected for this study will be shared with SomaLogic Inc., the company where sample testing and analysis will be done.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants 40 years and older
* Diagnosis of type 2 diabetes (T2D) [according to American Diabetes Association (ADA) guidelines]
* Able to provide consent
* Eligible for (per drug label/guidelines) at least one of the following drug classes: sodium-glucose cotransporter 2 inhibitors (SGLT2i), proprotein convertase subtilisin/kexin type 9 (PCSK9i), glucagon-like peptide receptor agonists (GLP-1 RA) but not currently prescribed any of these classes of drugs, or only prescribed PCSK9i

Exclusion Criteria:

* Systemic Lupus Erythematous (SLE)
* Pregnancy
* Intolerance or contraindication for use of GLP-1 RA, SGLT2i, and PCSK9i
* History of, an active, or untreated malignancy, in remission from a clinically significant malignancy (other than basal or squamous cell skin cancer, in situ carcinomas of the cervix, or in situ prostate cancer) for less than 5 years prior to, or are receiving or planning to receive therapy for cancer, at screening
* Inability to understand English (currently, SomaSignal testing information, guides, educational materials, and reports are only available in English.)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2022-02-03 (Actual); Primary Completion 2023-12-09 (Actual); Study Completion 2023-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arshed Quyyumi, MD, Principal Investigator — Emory University
Locations (5):
- United States (5):
  - Grady Health System, Atlanta, Georgia
  - Emory Hospital Midtown, Atlanta, Georgia
  - Emory Clinic, Emory University Hospital, Atlanta, Georgia
  - Emory Hospital, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
Researchers will share data after the completion of the trial and publications are completed. The research team will share de-identified data on patient demographics, outcomes, and SomaSignal Test Results.
Supporting Information: Study Protocol, SAP
Time Frame: Researchers will share data after completion of the trial and initial data are published.
Access Criteria: Data will be shared via secured data transfer

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Emory Healthcare System in Atlanta, Georgia, USA. Participant enrollment began February 03, 2022, and all follow-up was complete by December 9, 2023.
Period: Overall Study
Arm/Group | SomaSignal Informed Medical Management SSCVD | Standard of Care (Uninformed Arm)
Started | 73 | 70
Completed | 54 | 56
Not Completed | 19 | 14
Not completed — Lost to Follow-up | 9 | 3
Not completed — Withdrawal by Subject | 7 | 11
Not completed — Screen Failures | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SomaSignal Informed Medical Management SSCVD | Standard of Care (Uninformed Arm) | Total
Number analyzed (Participants) | 73 | 70 | 143
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 22 | 47
  >=65 years | 48 | 48 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.63 (10.16) | 67.66 (9.79) | 68.15 (9.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 32 | 67
  Male | 38 | 38 | 76
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 9 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 34 | 31 | 65
  White | 31 | 29 | 60
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 73 | 70 | 143

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Type 2 Diabetes (T2D) Who Had Prescription Changes in Concordance With SSCVD Results
Description: The number of participants with type 2 diabetes (T2D) who had changes in prescriptions aligned with SSCVD results at baseline will be reported for the informed group. For the uninformed group, this represents the number of participants who had prescription changes, even though the healthcare provider (HCP) was not informed of the results. SSCVD results from participants at both the baseline and 6-month periods will be provided to the study team during the 6-month study visit. Any recommendations made by physicians to participants, after these test results, will be collected. Medical records will be reviewed to assess any changes in treatment strategies.
Time Frame: 6 months and 12 months after baseline
Population: Participants with valid data who completed study visits.
Measure: Count of Participants; unit: Participants
Arm/Group | SomaSignal Informed Medical Management SSCVD | Standard of Care (Uninformed Arm)
Number analyzed (Participants) | 70 | 70
Participants
  Six months after baseline | 45 | 13
  Twelve months after baseline: number analyzed (Participants) | 54 | 56
  Twelve months after baseline | 8 | 35

2. Secondary Outcome: Number of Participants With Changes in the SSCVD Results
Description: During the baseline and follow-up visits, participants will have blood samples drawn for the SSCVD test.
Time Frame: Baseline and 6 months
Population: Participants with valid data who completed study visits.
Measure: Count of Participants; unit: Participants
Arm/Group | SomaSignal Informed Medical Management SSCVD | Standard of Care (Uninformed Arm)
Number analyzed (Participants) | 70 | 70
Participants
  Baseline: Low Risk | 6 | 6
  Baseline: Medium-Low Risk | 23 | 27
  Baseline: Medium-High Risk | 18 | 22
  Baseline: HIgh Risk | 23 | 15
  6 months: number analyzed (Participants) | 54 | 56
  6 months: Low Risk | 7 | 1
  6 months: Medium-Low Risk | 19 | 23
  6 months: Medium-High Risk | 13 | 16
  6 months: HIgh Risk | 15 | 16

3. Secondary Outcome: Changes in Low-density Lipoprotein (LDL)
Description: A blood sample to measure LDL will be drawn during the baseline and follow-up visits. Electronic medical records (EMR) will also be reviewed.
Time Frame: 6 months and 12 months
Population: Participants who completed study visits.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | SomaSignal Informed Medical Management SSCVD | Standard of Care (Uninformed Arm)
Number analyzed (Participants) | 70 | 70
mg/dL
  Six months after baseline | -30 (5) | -12 (8)
  Twelve months after baseline: number analyzed (Participants) | 54 | 56
  Twelve months after baseline | -45 (4) | 25 (6)

4. Secondary Outcome: Changes in High-density Lipoprotein (HDL)
Description: A blood sample to measure HDL will be drawn during the baseline and follow-up visits. EMR Records will also be reviewed
Time Frame: 6 months and 12 months
Population: Participants with valid data who completed study visits.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | SomaSignal Informed Medical Management SSCVD | Standard of Care (Uninformed Arm)
Number analyzed (Participants) | 70 | 70
mg/dL
  Six months after baseline | 5 (1.5) | 2 (2.0)
  Twelve months after baseline: number analyzed (Participants) | 54 | 56
  Twelve months after baseline | 8 (1.2) | 4 (2.5)

5. Secondary Outcome: Changes in Triglycerides (TG) Levels
Description: A blood sample to measure TG will be drawn during the baseline and follow-up visits. EMR Records will also be reviewed.
Time Frame: 6 months and 12 months
Population: Participants with valid data who completed the study visits.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | SomaSignal Informed Medical Management SSCVD | Standard of Care (Uninformed Arm)
Number analyzed (Participants) | 70 | 70
mg/dL
  Six months after baseline | -60 (5) | -15 (10)
  Twelve months after baseline: number analyzed (Participants) | 54 | 56
  Twelve months after baseline | -15 (2) | -45 (15)

6. Secondary Outcome: Changes in Glucose Levels
Description: A blood sample to measure glucose will be drawn during the baseline and follow-up visits. EMR records will also be reviewed.
Time Frame: 6 months and 12 months
Population: Participants with valid data who completed study visits.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | SomaSignal Informed Medical Management SSCVD | Standard of Care (Uninformed Arm)
Number analyzed (Participants) | 70 | 70
mg/dL
  Six months after baseline | -45 (4) | 10 (8)
  Twelve months after baseline: number analyzed (Participants) | 54 | 56
  Twelve months after baseline | -10 (8) | 35 (12)

7. Secondary Outcome: Changes in Glycated Hemoglobin Test (HbA1C)
Description: A blood sample to measure HbA1C will be drawn during the baseline and follow-up visits.
Time Frame: 6 months and 12 months
Population: Participants with valid data who completed study visits.
Measure: Mean (Standard Deviation); unit: percent of RBCs with glycated hemoglobin
Arm/Group | SomaSignal Informed Medical Management SSCVD | Standard of Care (Uninformed Arm)
Number analyzed (Participants) | 70 | 70
percent of RBCs with glycated hemoglobin
  Six months after baseline | -1.8 (1.3) | 0.8 (0.2)
  Twelve months after baseline: number analyzed (Participants) | 54 | 56
  Twelve months after baseline | -2.2 (1.2) | -2.4 (1)

8. Secondary Outcome: Changes in Weight
Description: Weight will be measured in kilograms (kg) during baseline and follow-up visits. EMR records will also be reviewed.
Time Frame: 6 months and 12 months
Population: Participants with valid data who completed study visits.
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | SomaSignal Informed Medical Management SSCVD | Standard of Care (Uninformed Arm)
Number analyzed (Participants) | 70 | 70
Kilograms
  Six months after baseline | -6.37 (0.4) | 0.87 (0.3)
  Twelve months after baseline: number analyzed (Participants) | 54 | 56
  Twelve months after baseline | -3.47 (0.2) | -3.18 (01)

9. Secondary Outcome: Changes in Body Mass Index (BMI)
Description: Height will be measured in meters (m) during the baseline visit, and weight will be measured during the baseline and follow-up visits. BMI will be calculated at each visit using the formula: weight (kg) / [height (m)]^2. EMR will also be reviewed.
Time Frame: 6 months and 12 months
Population: Participants with valid data who completed study visits.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | SomaSignal Informed Medical Management SSCVD | Standard of Care (Uninformed Arm)
Number analyzed (Participants) | 70 | 70
kg/m^2
  Six months after baseline | -2.2 (0.4) | 0.3 (0.2)
  12 months after baseline: number analyzed (Participants) | 54 | 56
  12 months after baseline | -1.2 (0.3) | 1.1 (0.1)

10. Secondary Outcome: Number of Participants Who Experienced Changes in Tobacco Exposure
Description: Participants will complete a questionnaire on personal tobacco use and exposure to second-hand smoke at both the baseline and follow-up visits. Responses are provided as categorical, multiple-choice options, and no summary score will be calculated for tobacco exposure. Data will also be extracted from the EMR.
Time Frame: 6 months and 12 months
Population: Participants with valid data who completed the study visit.
Measure: Count of Participants; unit: Participants
Arm/Group | SomaSignal Informed Medical Management SSCVD | Standard of Care (Uninformed Arm)
Number analyzed (Participants) | 70 | 70
Participants
  Six months after baseline | 3 | 1
  Twelve months after baseline: number analyzed (Participants) | 54 | 56
  Twelve months after baseline | 10 | 5

11. Secondary Outcome: Number of Participants Who Experienced a Change in Physical Activity
Description: A questionnaire will be provided at baseline and follow-up visit asking about physical activity habits. The questionnaire asks respondents how active they are during leisure time and has four response options:
  * Mainly sedentary (e.g. sitting, reading, watching television)
  * Mild exercise, minimal effort (eg. yoga, archery, sport fishing, easy walking at least 3 times per week)
  * Moderate exercise (eg. walking, bicycle riding, or light gardening at least 4 hours per week)
  * Strenuous exercise (heart beats rapidly e.g. running/jogging, football, vigorous swimming at least 3 times per week)
  A summary score is not calculated for this assessment. Data will also be extracted from EMR.
Time Frame: 6 months and 12 months
Population: Participants with valid data who completed the study visit.
Measure: Count of Participants; unit: Participants
Arm/Group | SomaSignal Informed Medical Management SSCVD | Standard of Care (Uninformed Arm)
Number analyzed (Participants) | 70 | 70
Participants
  Six month safter baseline | 25 | 3
  Twelve months after baseline: number analyzed (Participants) | 54 | 56
  Twelve months after baseline | 12 | 19

12. Secondary Outcome: Number of Participants Who Changed Their Dietary Habits
Description: Dietary habits will be assessed with a 5-item asking about consumption of salty foods, deep fried foods, fruits, vegetables, and meat/poultry. Responses are given as yes or no. There is not a summary score generated for this questionnaire.
Time Frame: 6 months and 12 months
Population: Participants with valid data who completed study visits.
Measure: Count of Participants; unit: Participants
Arm/Group | SomaSignal Informed Medical Management SSCVD | Standard of Care (Uninformed Arm)
Number analyzed (Participants) | 70 | 70
Participants
  Six months after baseline | 25 | 3
  Twelve months after baseline: number analyzed (Participants) | 54 | 56
  Twelve months after baseline | 12 | 19

13. Secondary Outcome: Physician Experience Questionnaire
Description: The physician questionnaire will ask 6 to 8 open ended and multiple choice questions regarding changes to treatment plans, identification of unexpected higher risk patients patients, and frequency of testing preferences. There is not a summary score generated for this qualitative questionnaire.
Time Frame: At 6 months
Population: This data was not collected on any of the participants
Arm/Group | SomaSignal Informed Medical Management SSCVD | Standard of Care (Uninformed Arm)
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Change in Medication Possession Ratio
Description: Participant adherence to medications will be quantified using the medication possession ratio which is the number of prescriptions filled divided by the number of months participants are prescription eligible.
Time Frame: Baseline and 6 months
Population: Data not collected
Arm/Group | SomaSignal Informed Medical Management SSCVD | Standard of Care (Uninformed Arm)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected from the time consent to participate in the study was given until 6 months after consent.
Arm/Group | SomaSignal Informed Medical Management SSCVD | Standard of Care (Uninformed Arm)
All-Cause Mortality (participants affected / at risk) | 0/73 | 0/70
Serious Adverse Events (participants affected / at risk) | 1/73 | 0/70
Other Adverse Events (participants affected / at risk) | 0/73 | 0/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SomaSignal Informed Medical Management SSCVD (N=73) | Standard of Care (Uninformed Arm) (N=70)
Non related hospital admission (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — The participant had low potassium on baseline research labs, was admitted with shortness of breath and tremors, treated for heart failure, repleted potassium, started SGLT2I at discharge, but discontinued due to urinary tract infection (UTI).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2022-11-14): https://cdn.clinicaltrials.gov/large-docs/06/NCT05256706/Prot_001.pdf